CLINICAL TRIAL: NCT02518399
Title: Chronic Heat Therapy for Improving Biomarkers of Vascular Health in Young, Healthy, Humans
Brief Title: Chronic Heat Therapy for Improving Vascular Health
Acronym: CHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Principal Investigator, Christopher T Minson, PhD, Professor, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09272013.025; 14PRE20380300 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2015-07-23; First posted 2015-08-07 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Diseases
Keywords: Blood vessels; Heat; Cardiovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heat therapy (Experimental): Subjects will report to the laboratory 4-5x per week for 8 weeks (36 sessions total) for heat therapy sessions. In each session, subjects will be immersed in a 40°C hot tub for up to 90min in order to increase body core temperature to 38.5°C and, once there, maintain it between 38.5-39.0°C for 60min.
  Interventions: Other: Heat therapy
- Thermoneutral water immersion (Sham Comparator): Subjects will report to the laboratory 4-5x per week for 8 weeks (36 sessions total) for thermoneutral water immersion sessions. In each session, subjects will be immersed in a 36°C tub for 90min in order to maintain body core temperature at a constant level.
  Interventions: Other: Thermoneutral water immersion

INTERVENTIONS:
Other: Heat therapy — Subjects will report to the laboratory 4-5x per week for 8 weeks (36 sessions total) for heat therapy sessions. In each session, subjects will be immersed in a 40°C hot tub for up to 90min in order to increase body core temperature to 38.5°C and, once there, maintain it between 38.5-39.0°C for 60min.
  Arms: Heat therapy
Other: Thermoneutral water immersion — Subjects will report to the laboratory 4-5x per week for 8 weeks (36 sessions total) for thermoneutral water immersion sessions. In each session, subjects will be immersed in a 36°C tub for 90min in order to maintain body core temperature at a constant level.
  Arms: Thermoneutral water immersion

SUMMARY:
The purpose of the study is to investigate whether long-term heat therapy (i.e. 8 weeks of hot tub 4-5x per week) improves biomarkers of cardiovascular health in young, healthy, able-bodied individuals. Although exercise is a potent means of improving cardiovascular health, many patients are unable to exercise effectively, and thus there is high demand for novel therapies to better manage cardiovascular risk in these patients. If successful, this study will set the groundwork for heat therapy to be used as an alternative treatment in patients who have limited exercise capabilities for the prevention of cardiovascular disease.

DETAILED DESCRIPTION:
Exercise training is a potent means of improving cardiovascular (CV) risk; however, exercise is challenging for many patient populations. Passive heat therapy may provide a simple and effective alternative to exercise for improving CV health, and no one has yet studied the physiological benefits of chronic heat exposure in humans. Heat exposure induces the expression of heat shock proteins, which can have a multitude of beneficial effects on the CV system, many of which are common to exercise training. In particular, these benefits include upregulation of many cellular pathways associated with improved vascular function, a predominant contributor to CV health. The goal of the study is to determine the effects of chronic passive heat therapy on vascular function in young, healthy, able-bodied individuals. The investigators will perform a randomized-controlled trial in which subjects participate in 8 weeks of either heat therapy or thermoneutral water immersion (sham). Heat therapy will entail 8 weeks of hot water immersion sufficient to raise core temperature >38.5°C for 1h, 4-5 times per week. Thermoneutral water immersion will entail 8 weeks of immersion in 36°C water for the same duration as heat therapy. In both subject groups, the investigators will measure various well-established biomarkers of vascular function before and after 8 weeks of heat therapy, including measures of arterial stiffness (arterial compliance, beta-stiffness, and pulse wave velocity), endothelium-dependent dilation (flow-mediated dilation), and intima media thickness. The investigators will investigate the effects of heat therapy on the microvasculature and on the mechanisms behind improvements in vascular function in the cutaneous microcirculation, an ideal site for pharmacodissecting the molecular pathways involved, using microdialysis paired with laser-Doppler flowmetry. If successful, these studies will serve as a basis for developing heat therapy as a novel means of improving CV risk, which has the potential to reshape the treatment of patient populations with limited exercise capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Young, healthy, able-bodied

Exclusion Criteria:

* Diagnosis of any chronic diseases related to the cardiovascular system (e.g. hypertension, cardiovascular disease, diabetes, etc.),
* Currently taking prescription medications (except contraceptives)
* Body mass index over 27 kg/m2
* Current smoking
* Currently pregnant or breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Change in flow-mediated dilation | 8 weeks
  The change in percent dilation of the brachial artery following release of a 5-min arterial occlusion, measured using ultrasonography. This test is highly prognostic of cardiovascular risk and mortality.
Femoral dynamic arterial compliance | 8 weeks
  The change in compliance of the superficial femoral artery relative to blood pressure, measured using ultrasonography-tonometry. This is a measure of arterial stiffness.
Intima media thickness | 8 weeks
  Change in wall thickness of the common carotid artery, measured using ultrasonography. This is predictive of future development of cardiovascular disease, in particular, atherosclerosis.
Mean arterial blood pressure | 8 weeks
  Change in blood pressure measured using brachial oscillation following >20 min supine rest.

SECONDARY OUTCOMES:
Cutaneous nitric oxide-dependent dilation | 8 weeks
  Change in the difference between cutaneous microdialysis sites receiving a nitric oxide inhibitor (L-NNA, IND # 124,303) and Lactated Ringer's (control). Measured using laser-Doppler flowmetry during a local heating protocol.

OTHER OUTCOMES:
Carotid dynamic arterial compliance | 8 weeks
  Change in compliance of the common carotid artery relative to blood pressure, measured using ultrasonography-tonometry. This is a measure of arterial stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

REFERENCES:
- [Result] Brunt VE, Howard MJ, Francisco MA, Ely BR, Minson CT. Passive heat therapy improves endothelial function, arterial stiffness and blood pressure in sedentary humans. J Physiol. 2016 Sep 15;594(18):5329-42. doi: 10.1113/JP272453. Epub 2016 Jun 30. PMID 27270841